CLINICAL TRIAL: NCT01367834
Title: Effect of Growth Hormone on Early Brain Development in Girls With Turner Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rebecca Knickmeyer Santelli, PhD (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor-Investigator, Rebecca Knickmeyer Santelli, PhD, Associate Professor, University of North Carolina, Chapel Hill
Organization: University of North Carolina, Chapel Hill (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 09-2171
Record Dates: First submitted 2011-06-02; First posted 2011-06-07 (Estimated); Results first posted 2017-03-24 (Actual); Last update posted 2017-03-24 (Actual); Status verified 2017-02

CONDITIONS: Turner Syndrome
Keywords: Turner Syndrome; growth hormone; brain development
MeSH Terms: conditions — Turner Syndrome | interventions — Growth Hormone; Human Growth Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Growth Hormone (Experimental): Subjects in the somatotropin (growth hormone, GH) arm will receive GH injections from 12-24 months of life.
  Interventions: Drug: somatotropin
- Control (No Intervention): Subjects will receive no GH or placebo.

INTERVENTIONS:
Drug: somatotropin — Subjects will receive 5 mg somatotropin (growth hormone) pens with cartridges. Subcutaneous injections are to be given every evening around bedtime. Dosing regimen: 50 mcg/kg/day to be adjusted at 4 month intervals to the closest 0.1 mg. Subjects will be given 12 months of treatment (from 12 to 24 months of life). Subjects will visit their pediatrician or pediatric endocrinologist at 4 and 8 months of life.
  Other Names: Genotropin; Growth hormone
  Arms: Growth Hormone

SUMMARY:
The purpose of this research study is to learn about brain development in very young girls with Turner syndrome (TS) and the effect that growth hormone (GH) therapy has on early brain development.

DETAILED DESCRIPTION:
Studies in older children and adults have found that IQ (intelligence quotient) in individuals with Turner syndrome (TS) and the general population are similar. However, many individuals with TS have a nonverbal learning disability which may cause problems with imagining and working with objects in space (for example: building blocks, working puzzles, copying designs, driving a car) as well as problems in planning, paying attention, and getting along with people their own age. Studies of brain structure have found changes in the size and function of specific areas of the brain that are involved in these nonverbal processes. However, there are no data published on brain structure or function in girls with Turner Syndrome in the first few years of life when brains are learning and growing most rapidly.

In a recent study, very young, short girls with Turner Syndrome (TS)(averaging 2 years in age) were treated with Growth Hormone (GH) and almost reached an average height after 2 years. The risks of GH for the young girls in that study appeared to be the same as those for older girls. Therefore, it is now recommended that GH therapy be considered as soon as a child with TS has growth failure. Growth failure often occurs during infancy; therefore, more children with TS are now receiving GH therapy as young as 12 months of age. In this study, the investigators wish to start understanding what effect GH has on learning and brain growth when given between the ages of 12 and 24 months. In this study, the girls with TS will have developmental studies, a physical examination, magnetic resonance imaging (MRI), and blood drawn at one and two years of age. Some of the girls in this study will receive GH from 12 until 24 months of life, while others will not. Brain growth and development will be compared between those who have been treated with GH and those who have not. This is a pilot study in which the investigators will gather data to design a larger study that can answer these questions.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Turner syndrome
* Less than the 50th percentile for length for the general female population

Exclusion Criteria:

* Prior Growth Hormone (GH) therapy
* Diabetes
* Allergy to metacresol (a preservative in the GH liquid that is injected)
* Contraindications for Magnetic Resonance Imaging (MRI) (such as metal in the body)
* Part of a Y chromosome in child's karyotype
* Parent/guardian is not willing for child to be randomized to be in the treatment group (receives Growth Hormone injections for one year) or the control group (receives no Growth Hormone during the study)
* Parent/guardian is not willing for child to have some of her developmental testing digitally recorded for scoring

Ages: 11 Months to 13 Months | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Enrollment: 17 (Actual)
Dates: Start 2010-05; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Knickmeyer, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited locally in the UNC_Chapel Hill pediatric endocrinology clinic and nationally through the Turner Syndrome Society, Turner Syndrome family internet groups, and advertisements on our UNC research website.
Groups:
- Growth Hormone: Subjects in the growth hormone (GH) arm will receive GH injections from 12-24 months of life.
  somatotropin: Subjects will receive 5 mg somatotropin (growth hormone) pens with cartridges. Subcutaneous injections are to be given every evening around bedtime. Dosing regimen: 50 mcg/kg/day to be adjusted at 4 month intervals to the closest 0.1 mg. Subjects will be given 12 months of treatment (from 12 to 24 months of life). Subjects will visit their pediatrician or pediatric endocrinologist at 4 and 8 months of life.
Period: Overall Study
Arm/Group | Growth Hormone | Control
Started | 11 | 6
Completed | 9 | 3
Not Completed | 2 | 3
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Study was ended. | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Growth Hormone | Control | Total
Number analyzed (Participants) | 11 | 6 | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 11 | 6 | 17
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: months] | 13.12 (0.82) | 12.73 (0.50) | 12.96 (0.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 6 | 17
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 11 | 6 | 17

OUTCOME MEASURES:

1. Primary Outcome: Total Brain Volume
Description: Percent change in total brain volume as determined by magnetic resonance imaging (MRI)
Time Frame: Change in volume from 12 months of age scan in 24 months of age scan
Population: Note that only subjects with usable MRI data are included in this analysis (this is a subset of all children completing the protocol).
Measure: Mean (Standard Deviation); unit: percentage change
Groups:
- Growth Hormone: Subjects in the growth hormone (GH) arm will receive GH injections from 12-24 months of life.
- Control: No intervention
Arm/Group | Growth Hormone | Control
Number analyzed (Participants) | 5 | 1
percentage change | 18.22 (1.99) | 19.78 (NA) — N of 1

2. Secondary Outcome: Volume of Brain Lobes (Occipital)
Description: Percent change in volumes of occipital lobes as determined by MRI.
Time Frame: Change in volume from 12 months of age scan in 24 months of age scan
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Growth Hormone | Control
Number analyzed (Participants) | 5 | 1
percentage change | 14.83 (2.21) | 12.16 (NA) — N = 1

3. Secondary Outcome: White Matter Tracts (SLF)
Description: Change in the fractional anisotropy (FA) of white matter tracts using Diffusion Tensor Imaging (DTI); superior longitudinal fasciculus
Time Frame: Change in FA from 12 months of age scan in 24 months of age scan
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Growth Hormone | Control
Number analyzed (Participants) | 4 | 1
percentage change | 15.12 (5.01) | 16.35 (NA) — N = 1

4. Secondary Outcome: Volume of Brain Lobes (Central)
Description: Percent change in volumes of central brain region (precentral gyrus, postcentral gyrus, rolandic operculum) as determined by MRI.
Time Frame: Change in volume from 12 months of age scan in 24 months of age scan
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Growth Hormone | Control
Number analyzed (Participants) | 5 | 1
percentage change | 17.63 (2.13) | 10.23 (NA) — N = 1

5. Secondary Outcome: Volume of Brain Lobes (Frontal)
Description: Percent change in volumes of frontal lobes as determined by MRI.
Time Frame: Change in volume from 12 months of age scan in 24 months of age scan
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Growth Hormone | Control
Number analyzed (Participants) | 5 | 1
percentage change | 15.43 (1.84) | 14.38 (NA) — N = 1

6. Secondary Outcome: Volume of Brain Lobes (Temporal)
Description: Percent change in volumes of temporal lobes as determined by MRI.
Time Frame: Change in volume from 12 months of age scan in 24 months of age scan
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Growth Hormone | Control
Number analyzed (Participants) | 5 | 1
percentage change | 10.79 (3.68) | 5.08 (NA) — N = 1

7. Secondary Outcome: Volume of Brain Lobes (Parietal)
Description: Percent change in volumes of parietal lobes as determined by MRI.
Time Frame: Change in volume from 12 months of age scan in 24 months of age scan
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Growth Hormone | Control
Number analyzed (Participants) | 5 | 1
percentage change | 18.86 (5.01) | 11.95 (NA) — N = 1

8. Secondary Outcome: Volume of Brain Lobes (Limbic)
Description: Percent change in volumes of parietal lobes as determined by MRI.
Time Frame: Change in volume from 12 months of age scan in 24 months of age scan
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Growth Hormone | Control
Number analyzed (Participants) | 5 | 1
percentage change | 15.43 (2.99) | 22.71 (NA) — N = 1

9. Secondary Outcome: Volume of Brain Lobes (Insular Cortex)
Description: Percent change in volumes of parietal lobes as determined by MRI.
Time Frame: Change in volume from 12 months of age scan in 24 months of age scan
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Growth Hormone | Control
Number analyzed (Participants) | 5 | 1
percentage change | 15.79 (2.11) | 19.78 (NA) — N = 1

ADVERSE EVENTS:
Time Frame: Baseline and 1 year
Arm/Group | Growth Hormone | Control
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/6
Other Adverse Events (participants affected / at risk) | 0/11 | 0/6

LIMITATIONS AND CAVEATS:
Low scan success rate and subject drop out resulted in small sample size (5 GH treated, 1 control).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less